CLINICAL TRIAL: NCT05848453
Title: A Phase 1, Double Blind, Randomized, Placebo-Controlled First in Human Study, to Assess the Safety, Tolerability and Pharmacokinetics of BAP5191 Following Topical Application of Repeat Doses in Healthy Adult Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of BAP5191 in Healthy Adults Following Topical Application of Repeat Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bacoba AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other); Swiss TPH, Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Screening
Other Study IDs: BAP5191-101
Record Dates: First submitted 2023-03-27; First posted 2023-05-08 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 1 mg/mL (0.1%) BAC6027 formulation; placebo
  Interventions: Drug: BAP5191
- Cohort 2 (Experimental): 5 mg/mL (0.5%) BAC6027 formulation; placebo
  Interventions: Drug: BAP5191
- Cohort 3 (Experimental): 10 mg/mL (1.0%) BAC6027 formulation; placebo
  Interventions: Drug: BAP5191

INTERVENTIONS:
Drug: BAP5191 — Placebo

SUMMARY:
All enrolled participants will be randomized to 3 cohorts with 8 participants each and will receive BAP5191 and placebo topically on a square of 121 cm2 each in the left and right scapula region daily for 28 days, with a 28-d safety follow-up.

The squares will be covered with a semi-occlusive patch. The doses will escalate from Cohort 1 to Cohort 2 to Cohort 3.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy adult participants,18 to 65 years of age.
* Women of childbearing potential (WOCBP) must agree to use a highly effective form of contraception, from at least 7 days prior to first administration to 28 days after last administration.
* Male participants with WOCBP partner must be willing to use condoms from first IMP application to 90 days after last application.
* Body Mass Index (BMI) between 18 and 29.9 kg/m2. Body weight must be greater than 50 kg.
* Clinical laboratory parameters, vital signs, pulse oximetry, and ECG within the reference range from population studies, or showing no clinically relevant deviations.

Key Exclusion Criteria:

* Chronic use of immunosuppressants within 3 years prior to the first administration of the study drug.
* History of prior leishmaniasis or extensive travel to endemic regions within 1 year prior to the first administration of the study drug.
* Presence or history of severe adverse reaction to any drug, or sensitivity to components of the study medication or to adhesive bandages or tape.
* Skin diseases, excessive hair, tattoos, pigmentation, scars or moles that could interfere with patch application and skin assessment at the site of application.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
General safety (number, frequency, severity, seriousness and duration of adverse events) | From day 0 to day 55
  Summarized statistics on adverse events will be reported under categories such as total adverse events, serious adverse events, treatment emerging adverse events.
Blood pressure from baseline | From day 0 to day 55
  Change of blood pressure from baseline. Systolic and diastolic blood pressure will be assessed.
Heart rate from baseline | From day 0 to day 55
  Change of pulse rate from baseline.
Respiratory rate from baseline | From day 0 to day 55
  Change of respiratory rate from baseline.
Temperature from baseline | From day 0 to day 55
  Change of tympanic temperature from baseline.
ECG parameters from baseline | From day 0 to day 55
  Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline.
Local skin tolerability: dermal response score | From day 0 to day 55
  Summarized statistics of tolerability assessment based on dermal response score and other effects score. The dermal response score ranges from score 0 (better, No evidence of irritation) to score 7 (worse, Strong reaction spreading beyond test site).
Local skin tolerability: other effects score | From day 0 to day 55
  Summarized statistics of tolerability assessment based on dermal response score and other effects score. The other effects score ranges from score 0 (better, None observed) to score 4 (worse, Glazing with fissures, Film of dried serous exudates covering all or part of the patch site, Small petechial erosions and/or scabs).

SECONDARY OUTCOMES:
Cmax of BAC6027 | during the procedure, day 0 - day 31
  Peak Plasma Concentration (Cmax) of BAC6027, if detectable.
Tmax of BAC6027 | during the procedure, day 0 - day 31
  Time to reach Cmax (Tmax), in case of plasma concentration determined.
AUC of BAC6027 | during the procedure, day 0 - day 31
  Area under the curve (AUC) of the plasma concentration determined.
AUC (0-t), of BAC6027 | during the procedure, day 0 - day 31
  Concentration from time zero to the last quantifiable concentration at time t, in case plasma concentration can be determined.
T1/2 of BAC6027 | during the procedure, day 0 - day 31
  The plasma elimination half-life, In case plasma concentration can be determined.
AUC (0-∞) of BAC6027 | during the procedure, day 0 - day 31
  The AUC of the plasma concentration from time zero to infinity with extrapolation of the terminal phase, In case plasma concentration can be determined.

OTHER OUTCOMES:
Histopathological findings of skin biopsies taken after completion of treatment on Day 31. | after the last PK sample collection, Day 31.
  Description of histopathological observations by application site and dose administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Universität Basel Departement Klinische Forschung Ambulantes Studienzentrum, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No